CLINICAL TRIAL: NCT03197688
Title: Multicenter, Retrospective Chart Review of First-time Opsumit® (Macitentan) Users in the United States
Brief Title: Retrospective Chart Review of First-time Opsumit® (Macitentan) Users in the United States
Acronym: OrPHeUS
Status: Completed | Type: Observational
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: AC-055-510
Record Dates: First submitted 2017-05-12; First posted 2017-06-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Notapplicable: Not applicable as non-interventional study
  Interventions: Other: Notapplicable

INTERVENTIONS:
Other: Notapplicable — Not applicable as non-interventional study

SUMMARY:
The Opsumit Users registry (OPUS; NCT02126943) was developed to characterize the safety profile of Opsumit and to describe clinical characteristics and outcomes of patients newly treated with Opsumit in the post-marketing setting. It is expected that the recruitment target of the OPUS registry cannot be achieved within the planned time period (5000 Opsumit new users by October 2018). The OrPHeUS study is designed to supplement the OPUS registry with retrospectively identified first-time Opsumit users in order to achieve the desired sample size.

ELIGIBILITY:
Inclusion Criteria:

* Patients who initiated Opsumit for the first time between 19 October 2013 and 31 December 2016 (inclusive)
* Patients whose medical charts are available for data collection

Exclusion Criteria:

* Patient participation in the OPUS registry
* Patient participation in any clinical trial involving Opsumit treatment or macitentan investigational product

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who initiated Opsumit for the first time between 19 October 2013 and 31 December 2016 (inclusive) are eligible for OrPHeUS (i.e., eligibility period).
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Estimation of incidence rates of adverse events | Observation period from 19 Oct 2013 to 31 March 2017, Data collection from 1 Apr 2017 to 30 Jun 2018
  Incidence rates of liver test abnormalities, Occurrence of Hepatic Adverse Events (HAEs), Occurrence of any other Adverse Event (AE), Occurrence and reason for discontinuation of Opsumit treatment, hospitalization and death

SECONDARY OUTCOMES:
Description of demographic characteristics of patients | Observation period from 19 Oct 2013 to 31 March 2017, Data collection from 1 Apr 2017 to 30 Jun 2018
  To describe demographic characteristics of patients treated with Opsumit at beginning and during study time period
Description of clinical characteristics of patients | Observation period from 19 Oct 2013 to 31 March 2017, Data collection from 1 Apr 2017 to 30 Jun 2018
  To describe clinical characteristics of patients treated with Opsumit at beginning and during study time period

CONTACTS AND LOCATIONS:
Locations (106):
- United States (105):
  - Pulmonary Associates, Phoenix, Arizona
  - Cardiovascular Consultants, Phoenix, Arizona
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - David Geffen School of Medicine at University of California Los Angeles, Los Angeles, California
  - UCSF School of Medicine, San Francisco, California
  - Paloma Medical Group, San Juan Capistrano, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - University of Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Bay Area Cardiology Associates, Brandon, Florida
  - Florida Lung, Asthma and Sleep Specialists, Celebration, Florida
  - Frank Hull, MD, PA, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - West Pasco Pulmonary Associates, Hudson, Florida
  - Saint Vincent's Medical Center, Jacksonville, Florida
  - Medical Research of Central Florida, Leesburg, Florida
  - Independent Lung Associates, Melbourne, Florida
  - University of Miami, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Central Florida Pulmonary Group, P.A. - Downtown Orlando Office, Orlando, Florida
  - Bassetti Medical Research Inc, Sebring, Florida
  - Cardiovascular Medicine Associates, South Miami, Florida
  - Coastal Pulmonary and Critical Care, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida Hospital, Weston, Florida
  - Florida Medical Clinic, Zephyrhills, Florida
  - Piedmont Healthcare, Austell, Georgia
  - Southeastern Cardiology Associates, Columbus, Georgia
  - Wellstar Marietta Pulmonary Medicine, Marietta, Georgia
  - Bingham Memorial Hospital, Shelley, Idaho
  - Northwestern University, Chicago, Illinois
  - IU Health Physicians Pulmonary & Critical Care, Carmel, Indiana
  - Lutheran Hospital, Fort Wayne, Indiana
  - Indiana Internal Medicine Consultants, Greenwood, Indiana
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - CIC Associates, Clive, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The University of Kansas Physicians, Kansas City, Kansas
  - St. Elizabeth Healthcare Clinical Research Institute, Erlanger, Kentucky
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Pulmonary & Critical Care Specialists, Shreveport, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Beaumont Medical Center, Troy, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis University, St Louis, Missouri
  - Pulmonary Consultants Inc-St. Louis, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Pulmonary Specialties, LLC, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Barnabas Health Ambulatory Care Center, Newark, New Jersey
  - Pulmonary and Critical Care Associates, Union, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Pulmonary Health Physicians, Fayetteville, New York
  - Stony Brook University Hospital, Hauppauge, New York
  - Temple University Hospital, Middletown, New York
  - Winthrop University Hospital, Clinical Trials Center, Mineola, New York
  - Mount Sinai, New York, New York
  - Montefiore Medical Center - Bronx, The Bronx, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Mount Carmel Medical Group, Columbus, Ohio
  - Midwest Pulmonary & Sleep Research, Dayton, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - The University of Toledo Medical Center, Toledo, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Legacy Research Institute, Portland, Oregon
  - The Oregon Clinic, Portland, Oregon
  - Doylestown Health Cardiology, a division of Doylestown Health Physicians, Doylestown, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - AnMed Health Medical Center, Anderson, South Carolina
  - Carolina Cardiology Associates, Rock Hill, South Carolina
  - Sioux Falls Cardiovascular PC, Sioux Falls, South Dakota
  - Memorial Research Center, Chattanooga, Tennessee
  - Mid-South Pulmonary Specialists, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Premier Pulmonary CC and Sleep Medicine, PA, Denison, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Baylor Regional Medical Center at Plano, Plano, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Washington, Seattle, Washington
  - Spokane Respiratory Consultants, Spokane, Washington
  - Cardiac Study Center, Tacoma, Washington
  - Aurora Health Care - Saint Luke's Medical Center, Milwaukee, Wisconsin
- CardioPulmonary Research Center, Guaynabo, Puerto Rico

REFERENCES:
- [Derived] Melendres-Groves LD, Channick RN, Chin KM, McLaughlin VV, MacDonald G, Martin N, Ong R, Sandros M, Kim NH. Characteristics, Treatment Patterns and Outcomes of Patients with Pulmonary Arterial Hypertension by Race and Ethnicity Using Real-World Data from the Combined OPUS/OrPHeUS Studies. Adv Ther. 2025 Nov 19. doi: 10.1007/s12325-025-03403-4. Online ahead of print. PMID 41258625
- [Derived] Kim NH, Chin KM, McLaughlin VV, Ong R, MacDonald G, Martin N, Senatore A, Channick R. Macitentan and Tadalafil Combination Therapy in Patients with Pulmonary Arterial Hypertension and Cardiovascular Comorbidities: Real-World Evidence from OPUS and OrPHeUS. Adv Ther. 2025 Jul;42(7):3306-3333. doi: 10.1007/s12325-025-03180-0. Epub 2025 May 19. PMID 40388087
- [Derived] Chin KM, Channick R, Kim NH, Ong R, Turricchia S, Martin N, Mitchell L, McLaughlin VV. Macitentan in Pulmonary Arterial Hypertension Due to Congenital Heart Disease (CHD-PAH): Real-World Evidence from the OPUS/OrPHeUS Studies. Cardiol Ther. 2024 Dec;13(4):775-796. doi: 10.1007/s40119-024-00386-1. Epub 2024 Nov 25. PMID 39585521
- [Derived] Channick R, Chin KM, McLaughlin VV, Lammi MR, Zamanian RT, Turricchia S, Ong R, Mitchell L, Kim NH. Macitentan in Pulmonary Arterial Hypertension Associated with Connective Tissue Disease (CTD-PAH): Real-World Evidence from the Combined OPUS/OrPHeUS Dataset. Cardiol Ther. 2024 Jun;13(2):315-339. doi: 10.1007/s40119-024-00361-w. Epub 2024 Mar 7. PMID 38451426
- [Derived] Kim NH, Chin KM, McLaughlin VV, DuBrock H, Restrepo-Jaramillo R, Safdar Z, MacDonald G, Martin N, Rosenberg D, Solonets M, Channick R. Safety of Macitentan for the Treatment of Portopulmonary Hypertension: Real-World Evidence from the Combined OPUS/OrPHeUS Studies. Pulm Ther. 2024 Mar;10(1):85-107. doi: 10.1007/s41030-023-00251-x. Epub 2024 Jan 7. PMID 38184507